CLINICAL TRIAL: NCT05004467
Title: Clinical Predictive Effects of Mulligan Treatment in Patients With Chronic Neck Pain: a Machine Learning Approach
Brief Title: Clinical Predictive Effects of Mulligan Treatment in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Eleuterio Atanasio Sánchez Romero, Professor / Researcher, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clinical predictive effects
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Orthopedic Disorder of Spine; Placebo Effect; Disability Physical
Keywords: Therapeutic Effect; Manual Therapy; Physiotherapy; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Study design:
  A randomized, longitudinal, experimental, prospective, parallel and double-blind clinical trial will be carried out in which both the study subject and the researcher who made the measurements do not know which treatment group they belong to.
  Participants The sample was composed of 42 healthy patients residing in the Community of Madrid, all of whom were personally recruited for the study. All of them will have two different manual therapy techniques (Mulligan and placebo) for acute or subactute neck pain. All patients will read the information sheet that explains what the study will consist of, as well as the informed consent form, which they will voluntarily sign before the intervention.
  Each group will be given a different sentence: one group will attempt to influence with a positive expectation, another with a neutral expectation, and yet another will attempt to influence with a negative expectation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the subjects assigned to the groups nor the researchers who measured the variables knew which group they belonged to.
  Patients will be randomly assigned through GraphPad Software's QuickCals application (La Joya, CA, USA) to one of the 2 study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement technique (Experimental): The therapist applies supported pressure on right and left side and articular planes. Meanwhile, the patient executes active movements and the therapist is trying to find the specifies cervical joint to get partial or total painful relief or movements with restrictions.
  If the therapist couldn´t relief or remove pain or restriction with the pressure permorfem, he will readjust pressure and slide in differents planes of motion. It is necessary achieve that aim.
  After that, the patient stay in sit down raised position on a stool, with his back in contact with the wall.
  Hip, knee and ankle of the patient suppor a certain position: 90º of flexion which will be checked with a conventional goniometer. His hands are on the thighs. The treatment lasts 5 minutes.
  Interventions: Other: Mobilization With Movement Technique
- Placebo technique (Sham Comparator): Placebo manual technique is performed similar to experimental group technique but no slides are performed. The therapist simply embraces cervical region with boths hands, avoiding any pressure or any painfully caoture.
  Interventions: Other: Mobilization With Movement Technique

INTERVENTIONS:
Other: Mobilization With Movement Technique — The researcher explains cervical movements to the patient to be done while the technique is performed. This movements will be the painful and limited movements detected in goniometric intervention before the treatment and movements done actively and in all range of motion.

SUMMARY:
The aim of the study is the measurement and comparison of two manual therapy techniques, the Mulligan´s mobilization with movement technique, and de placebo technique, both applicated in patients with subacute neck pain.

DETAILED DESCRIPTION:
Study design:

A randomized, longitudinal, experimental, prospective, parallel and double-blind clinical trial was conducted, where both the study subject and the researcher performing the measurements do not know which treatment group they belong to. Patients were randomly assigned using GraphPad Software's QuickCals application (La Joya, CA, USA) to one of the 2 study groups: experimental group and placebo group.

Participants:

The sample was composed of 42 sub-acute and inespecific neck pain patients residing in the Community of Madrid, all of whom were recruited personally for the study. Experimental group includes 21 subjects who received a manual theraphy technique named Mobilization with Movement (MWM) for a total of four sessions, distributed in two sessions per week. . Placebo group includes 21 subjects who received a placebo technique the same times.

Measurement instruments:

The primary outcomes of interest were true and total cervical ROM, Pain Pressure Threshold (PPT), pain intensity, Neck Disabilty Index, anxiety scale and depression scale. Secondary outcomes were pain and/or neck stiffnes for musculosketletal causes.

Goniometry

This is the measurement of angles on the arc of motion of a joint. Goniometry is a quantitative variable and numerical and unit of measurement is in degrees.

Measurement of cervical motion was performed with the device CROM (Cervical Range Of Motion) due to the extensive evidence as to its reliability. This device has two gravity goniometers, indicating the mobility in the sagittal and frontal planes (measurement of the flexion-extension and lateral inclination, respectively). For the transverse plane, the goniometer has a compass, a magnet with magnetic resting on the shoulders to measure neck rotation.

Algometry

Consists in measuring the pain threshold pressure, by stimulating the receptors of pressure. This threshold is defined as the minimal amount of pressure that produces pain.

Algometry is a quantitative variable and gives numerical values in Kilograms/cm2.

To study algometry has relied on a digital algometer Wagner Force One Digital Force Gage FDX model 100 with an 1cm2 head. This device, used with a gradually application of manual force and consistently, and prior familiarity with the user, has a high fiability.

* Intensity of pain measured by visual analogue scale (VAS) just before and immediately after treatment.
* Neck disability index: Scale completed by the patient before tratment
* BECK: Scale completed by the patient before tratment.
* STAI: Scale completed by the patient before tratment.
* Mobilization with movement technique: Technique therapy applied to the experimental group.

Procedural protocol:

Measures were collected before and after intervention, stablishing the hypotesys about reasons and inmediate effects in relation with the tecnique applied.

No follows-up will be done to the patients. It is supposed like a bounding factor in that study.

- Goniometric measurements procedure: The patient position for goniometric measurement is similar to the physiotherapist intervention, described previously.

The patient actively and in all range of motion , perform flexion, extension, bilateral lateral flexion and bilateral rotation movements. And then, the therapist will gather the parameters at the end of every movement.

All goniometric measures will be reported three times and the average of three measurements will be calculated.

Goniometric informacion is collected just before the therapeutic intervention and five minutes later.

- Pressure algometer measurements procedure: The patient supine with algometer perpendicular to the exactly point for evaluation, and the pressure is increasing slowly and linearly. The intervention speed applied will be 1kg/cm2/second until the patient feels pain. Just in that moment, the researcher stops pressure.

Hereby a target response is favored due to fact that patient has more reaction time when he starts to feel pain. In that moment, the researcher interrumps exercised pressure with the algometer.

In every anatomical reference, three measures will be performed consecutively in intervals of 30 seconds for measurement to generate an average, neccesary for statical analysis.

Pain pressure threshold measure is performed just before therapeutic intervention and 5 minutes later.

- Anatomical References to study: Bilateral measurement of superior cervical region in spine C2: To plan a horizontal line between spine C2 to both sides, separated 1 cm to the spine point.

Bilateral measurement of superior cervical region in spine C7: To plan a horizontal line between spine C7 to both sides, separated 1cm to the spine point.

Superior Trapezius measurement: Horizontal line between acromion to spine C7 Lateral Epycondile measurement: lateral prominence of distal humeral epiphysis with the superior extremity supported on the table.

The algometer technique is performed just before therapeutic intervention and 5 minutes later.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 60 years.
* Neck pain with/without pain in upper limb/s.
* NDI ≥ 10
* Acceptance of the study and completion of the informed consent form.

Exclusion Criteria:

* Presenting physician-diagnosed "red flag" of non-musculoskeletal origin.
* Having had a Whiplash in the last 2 years.
* Use of cervical collar in the last year.
* Evidence of CNS involvement.
* Vestibular Disorders
* Inflammatory joint disease
* Spinal cord pathology
* Bone disease or marked osteoporosis
* Intervertebral disc protrusion
* Subjects who have received physiotherapeutic treatment of the cervical or thoracic region three months previously.
* Fractures, sprain or dislocation of the neck, occurred in a period of less than two months.
* Previous shoulder, upper limb and cervical spine surgery, which occurred in the twelve months prior to the investigation.
* Pregnancy
* Illness
* Voluntary abandonment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from base line and immediately after the intervention
  To evaluate the pain that the patient has, we use the VAS (Appendix 1). This is a 100 mm line that measures pain intensity. The left end of the line represents the absence of pain, while the right end represents the worst pain imaginable. The numerical pain intensity scale adds a numerical graduation where 1 is no pain and 10 is the worst pain imaginable. The confidence and reliability of this scale has been approved and validated in different studies. This scale will be used accompanying each CROM measurement as well as in pre-treatment measurements.
Pressure Pain Threshold | Change from base line and immediately after the intervention
  The patient supine with algometer perpendicular to the exactly point for evaluation, and the pressure is increasing slowly and linearly. The intervention speed applied will be 1kg/cm2/second until the patient feels pain. Just in that moment, the researcher stops pressure.
  Hereby a target response is favored due to fact that patient has more reaction time when he starts to feel pain. In that moment, the researcher interrumps exercised pressure with the algometer.
  In every anatomical reference, three measures will be performed consecutively in intervals of 30 seconds for measurement to generate an average, neccesary for statical analysis.
  Pain pressure threshold measure is performed just before therapeutic intervention and 5 minutes later.
Cervical Range of Movement (CROM) | Change from base line and immediately after the intervention
  Measurement of the range of movement by means of an inclinometer. To measure the range of movement the patient will be seated in a chair; feet supported on the floor, triple flexion of lower limbs of 90º (hip, knee and foot), back well supported and straight, head straight and look at the horizon. The inclinometer will be positioned to measure flexion, extension, right and left tilt and right and left rotation. The inclinometer for CROM (cervical range of motion) is approved and validated in different studies.

SECONDARY OUTCOMES:
Neck Disability Index | Change from base line and immediately after the intervention
  It will be used to measure the level of disability perceived by the patient as a result of their neck pain, after performing the technique and to check whether it appears during the control measurements. It is a questionnaire composed of 10 sections on different activities of daily living (ADLs); self-care, reading, lifting weights, driving, sleeping, recreational activities, work, concentration, pain intensity and headache. Each section scores from 0 to 5, with zero being no pain and five being the worst pain imaginable. (Maximum 50 points). Therefore, in order of appearance, of the 6 options, the first option of each item represents 0 and the last one 5. The higher the score obtained, the greater the patient's disability.
STAI (State-Trait Anxiety) | Change from base line and immediately after the intervention
  Questionnaire composed of 20 items with 4 points each that evaluate "state anxiety" (transitory emotional condition influenced by environmental factors that decrease or increase anxiety) and another 20 that evaluate "trait anxiety" (personality factor that predisposes to suffer or not suffer anxiety). The 2-part score ranks patients at a percentile to the general population. The higher the score, the greater the anxiety. It is one of the most widely used tools in research to measure levels of general anxiety.
Beck II (Depression) | Change from base line and immediately after the intervention
  A 21-item scale used to assess the severity of depression. The patient has to select for each item the response alternative that best reflects his/her state during the last week. The total score is obtained by adding up the values of the selected items, which range from 0 to 3. The commonly accepted cut-off points for grading intensity/severity are as follows: 0 to 9, no depression; 10 to 18, mild depression; 19 to 29, moderate depression, and ≥ 30 points, severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Study Director — Universidad Rey Juan Carlos; Eleuterio A Sánchez Romero, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Spain